CLINICAL TRIAL: NCT03912662
Title: Poetry Study - ProGrip™ Self-gripping Polyester Mesh Prospective Embedded REgisTRY for Abdominal Wall Sutureline Reinforcement in Subjects Undergoing Midline Laparotomy to Prevent Incisional Hernia
Brief Title: ProGripTM Self-Gripping Polyester Mesh in Incisional Hernia Prevention
Acronym: POETRY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Surgical complications arose early in the study, mainly due to patient complexity, not to study device or implantation. Despite refining protocol to exclude highly complex patients, these issues persisted, leading to the study's early termination.
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT17048POETRY
Record Dates: First submitted 2019-03-21; First posted 2019-04-11 (Actual); Results first posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Incisional Hernia
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hernia prevention cohort (Other): single arm safety study, no control arm
  Interventions: Device: Mesh augmented reinforcement

INTERVENTIONS:
Device: Mesh augmented reinforcement — Abdominal wall sutureline reinforcement with ProgripTM Self-Gripping Polyester Mesh

SUMMARY:
Interventional, prospective, multicenter, post-marketing clinical follow-up study.

After midline laparotomy, the probability to develop an incisional hernia ranges from 10% to 50% depending on the complexity of the surgery and patient state of health.

As the clinical data needed for the study corresponds with those collected by Club Hernie registry, the clinical study will use the established registry database to collect performance and safety data on the prevention of incisional hernias within 24 months post operatively.

DETAILED DESCRIPTION:
The primary objective of this investigation is to confirm the efficacy of ProGrip™ Self-gripping Polyester Mesh to reduce the incidence of incisional hernia within 24 months post-operatively in subjects undergoing procedures with midline laparotomies.

Secondary Objective The secondary objective of this investigation is to confirm the safety of ProGrip™ Self-gripping Polyester Mesh through the occurrence of adverse device effects or procedure related adverse events following the use of ProGrip™ Self- gripping Polyester Mesh in subjects undergoing procedures with midline laparotomies.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided informed consent.
2. Subject is ≥ 18 years of age at the time of consent.
3. Subject will be undergoing an elective midline laparotomy.
4. Subject may have a combination of low- and high-risk factors but cannot exceed a total of 5 risk factors or have more than 2 high-risk factors. Subject must have at least 2 low-risk factors if subject does not have any high-risk factors. High- and low-risk factors include:

   1. High-Risk Factors (maximum of 2): i.BMI≥ 35; ii.Prior open abdominal surgery; iii.Daily active smoker or Chronic Obstructive Pulmonary disease (COPD) diagnosis; iv. Current or recent (within 1 year) cancer diagnosis or chemotherapy treatment; v.History of or current abdominal aorta aneurism or surgery for abdominal aortaaneurism
   2. Low-Risk Factors (minimum of 2, if no high-risk factors): i.25 ≤ BMI < 35; ii.Age > 45; iii.Uncontrolled diabetes; iv.Malnutrition as defined by 10% weight loss within the last 3 months; v.Current immunosuppressive treatment; vi.Undergoing colorectal surgery

Exclusion Criteria:

1. Subject is undergoing emergency surgery, i.e. lifesaving procedures performed where subject is in imminent danger of death.
2. Subject for which the device is used outside the product IFU, including;

   1. Pregnant women: Women who are known or suspected to be pregnant, or who are planning to become pregnant during the study follow-up period
   2. Subject who has an infection within 30 days of enrollment or, at the time of the surgery, has any active, acute or chronic infection(s) that are uncontrolled and/or requiring treatment such as antibiotics
   3. Subject whose surgical site is contaminated or dirty/infected intraoperatively, as assessed by the Investigator (Exclude Altemeier classification III-IV).
3. Subject who had received a mesh in a previous ventral hernia repair or has a ventral hernia.
4. Investigator determined that a planned future surgery would interfere with application of mesh reinforcement.
5. Subject has participated in an investigational drug or device research study within 30 days of enrollment.
6. Subject has a life expectancy of <2 years.
7. Subject has an ASA Physical Status Classification System score >3.
8. Subject has >5 total risk factors or >2 high-risk factors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Bertrand, MD, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (11):
- France (11):
  - CHU Besançon, Besançon
  - CHU de Bordeaux, Bordeaux
  - CHU de Bordeaux - Hôpital Haut-Lévêque, Bordeaux
  - CHU Lille, Lille
  - HCL Louis Pradel, Lyon
  - CHU de Nantes, Nantes
  - CHU de Nîmes, Nîmes
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - CHU Hopitaux de Rouen, Rouen
  - CHU Strasbourg - Nouvel Hôpital Civil, Strasbourg

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A subject is considered enrolled in the study when it is confirmed they meet all pre-operative inclusion and no exclusion criteria, the Informed Consent Form is signed and they have been implanted with the device.
Groups:
- Patients Consented for POETRY Study: Patients consented for POETRY Study and may recieve ProGrip™ Self-Gripping Polyester Mesh.
Period: Overall Study
Arm/Group | Patients Consented for POETRY Study
Started (There were 35 screened and consented subjects.) | 35
Enrolled (Received Study Device) (Consented subjects who meet all pre-operative inclusion and no exclusion criteria, and have been implanted with the device.) | 32
Safety Analysis Set | 32
Completed | 6
Not Completed | 29
Not completed — Adverse Event | 3
Not completed — Adverse Event and Death | 1
Not completed — Death | 1
Not completed — Screen Failure: Subjects who provide study consent, but then were determined to be ineligible. | 1
Not completed — Mesh Removal | 1
Not completed — Discontinued: Eligible consented subjects who did not undergo the procedure with the study device. | 2
Not completed — Early study termination | 20

BASELINE CHARACTERISTICS:
Groups:
- Patients Treated With ProGrip™ Self-Gripping Polyester Mesh: ProGrip™ Self-Gripping Polyester Mesh: All subjects enrolled who received the ProGrip™ Self-Gripping Polyester Mesh
Arm/Group | Patients Treated With ProGrip™ Self-Gripping Polyester Mesh
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (13.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Mean (Standard Deviation); unit: kg] | 73.6 (17.96)
Height [Mean (Standard Deviation); unit: cm] | 169.5 (9.26)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.5 (5.66)
Work [Count of Participants; unit: Participants]
  Unemployed | 16
  Administrative work | 4
  Moderately physical labor | 5
  Physical labor | 3
  Not Provided | 4
Sport Activity [Count of Participants; unit: Participants]
  None | 14
  Intense (>1x/week) | 3
  Moderate (1x/week) | 14
  Sporadic | 1

OUTCOME MEASURES:

1. Primary Outcome: Incisional Hernia Rate
Description: Incisional hernia rate within 24 months of midline laparotomy assessed by CT-scan and physical examination including hernia clinical examination.
Time Frame: 24 months
Population: Patients who received ProGrip Self-Gripping Polyester Mesh for suture line reinforcement after midline laparotomy, met all of the inclusion criteria, and none of the exclusion criteria.
Measure: Count of Participants; unit: Participants
Groups:
- Patients Treated With ProGrip Self-Gripping Polyester Mesh and 24-Months of Study Follow-up: Four patients who received the ProGrip Self-Gripping Polyester Mesh and who completed the 24-month visit.
Arm/Group | Patients Treated With ProGrip Self-Gripping Polyester Mesh and 24-Months of Study Follow-up
Number analyzed (Participants) | 4
Participants | 1

2. Secondary Outcome: Adverse Event
Description: AE incidence reported by number, seriousness, and relationship to the procedure and device from the surgery to the 24-month visit
Time Frame: From the surgery to the 24-month visit
Population: as for outcome 1
Measure: Number; unit: Adverse Events
Groups:
- Patients Treated With ProGrip™ Self-Gripping Polyester Mesh: ProGrip™ Self-Gripping Polyester Mesh: All subjects enrolled receiving the ProGrip™ Self-Gripping Polyester Mesh
Arm/Group | Patients Treated With ProGrip™ Self-Gripping Polyester Mesh
Number analyzed (Participants) | 32
Adverse Events
  Total Number of Adverse Events | 39
  Number of SAEs | 25
  Number of non-Serious AEs | 14
  Number of Device-Related AEs | 8
  Number of Mesh Placement Procedure-related AEs | 5
  Number of Device-related SAEs | 6
  Number of Mesh Placement Procedure-related SAEs | 3
  Number of Index Procedure related AEs | 27
  Number of Index Procedure related SAEs | 14
  Number of AEs with action taken | 38
  AEs by reason for Seriousness: Hospitalization | 18
  AEs by reason for Seriousness: Death | 2
  AEs by reason for Seriousness: Life threatening illness or injury | 8
  AEs by reason for Seriousness: Permanent impairment of a body structure or body function | 1
  AEs by reason for Seriousness: Medical or surgical intervention | 19
  AEs by Relation to Study Device: Not Related | 31
  AEs by Relation to Study Device: Related | 8
  AEs by Relation to Index Procedure: Not Related | 12
  AEs by Relation to Index Procedure: Related | 27
  AEs by Relation to Mesh Placement Procedure: Not Related | 24
  AEs by Relation to Mesh Placement Procedure: Related | 4

3. Secondary Outcome: Time to Incisional Hernia Occurrence
Description: Time to incisional hernia occurrence from the surgery to the 24-month visit
Time Frame: From the surgery to the 24-month visit
Population: as for outcome 1
Measure: Median (Full Range); unit: Days to hernia occurrence
Groups:
- Patients Treated With ProGrip Self- Gripping Polyester Mesh: ProGrip™ Self-Gripping Polyester Mesh: All subjects enrolled receiving the ProGrip™ Self-Gripping Polyester Mesh
Arm/Group | Patients Treated With ProGrip Self- Gripping Polyester Mesh
Number analyzed (Participants) | 32
Days to hernia occurrence | 384 [384 to 384]

4. Secondary Outcome: Post-operative Pain at the Site of Surgery
Description: Post-operative pain at the site of the surgery was measured at days 0, 1, 8 and months 1, 12, 24 using a Visual Analog Scale - a psychometric response scale (0-10) (0 no pain, 10 the worst) either during systematic clinical visit or by phone call when a subject is already discharged. (Worst pain experienced over the last 24 hours).
Time Frame: Day 0, Day 1, Day 8, Month 1, Month 12, Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale of 0-10
Arm/Group | Patients Treated With ProGrip™ Self-Gripping Polyester Mesh
Number analyzed (Participants) | 30
score on a scale of 0-10
  EVA (VAS) Day 0 | 3.8 (2.94)
  EVA (VAS) Day 1 | 3.7 (2.73)
  EVA (VAS) Day 8: number analyzed (Participants) | 29
  EVA (VAS) Day 8 | 1.9 (2.42)
  EVA (VAS) Month 1: number analyzed (Participants) | 25
  EVA (VAS) Month 1 | 0.4 (0.91)
  EVA (VAS) Month 12: number analyzed (Participants) | 15
  EVA (VAS) Month 12 | 0.5 (1.81)
  EVA (VAS) Month 24: number analyzed (Participants) | 4
  EVA (VAS) Month 24 | 0 (0)

5. Secondary Outcome: Quality of Life Questionnaire (QOL) for Patient
Description: Assessment with Club Hernie Registry QOL questionnaire of patients treated with ProGrip Self-Gripping Polyester Mesh for suture line mesh reinforcement. . Two sets of self-administered QOL were administered; one for 1 month and one for 12- and 24-month.
Time Frame: Month 1, Month 12, Month 24
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Patients Treated With ProGrip™ Self-Gripping Polyester Mesh
Number analyzed (Participants) | 25
participants
  Month 1 : Post-operative discomfort: No symptoms | 16
  Month 1 : Post-operative discomfort: Discomfort | 3
  Month 1: Post-operative discomfort: Tingling (dyesthesia, hyperesthesia, hyperpathia) | 1
  Month 1: Post-operative discomfort: Reduced sensitivity | 3
  Month 1: Post-operative discomfort: Moderated pain per Visual Analog Scale (VAS) | 3
  Month 1: Post-operative discomfort: Other symptoms | 3
  Month 1: Post-operative discomfort: Response missing | 8
  Month 12 : Post-operative discomfort: No symptoms: number analyzed (Participants) | 16
  Month 12 : Post-operative discomfort: No symptoms | 14
  Month 12: Post-operative discomfort: Significant pain: number analyzed (Participants) | 16
  Month 12: Post-operative discomfort: Significant pain | 1
  Month 12: Post-operative discomfort: Other symptoms: number analyzed (Participants) | 16
  Month 12: Post-operative discomfort: Other symptoms | 1
  Month 24 : Post-operative discomfort: No symptoms: number analyzed (Participants) | 4
  Month 24 : Post-operative discomfort: No symptoms | 3
  Month 24: Post-operative discomfort: Reduced sensitivity: number analyzed (Participants) | 4
  Month 24: Post-operative discomfort: Reduced sensitivity | 1
  Month 1: Location of symptoms: Not applicable | 17
  Month 1: Location of symptoms: Side operated on | 6
  Month 1: Location of symptoms: Contralateral | 2
  Month 1: Location of symptoms: Elsewhere | 2
  Month 1: Location of symptoms: Response missing | 7
  Month 1: Timing of symptoms: Not applicable | 19
  Month 1: Timing of symptoms: after exertion or end of day | 3
  Month 1: Timing of symptoms: Anytime | 2
  Month 1: Timing of symptoms: During other activities | 2
  Month 1: Timing of symptoms: Response missing | 7
  Month 1: Frequency of symptoms: Not applicable | 19
  Month 1: Frequency of symptoms: Several times per day | 1
  Month 1: Frequency of symptoms: Often during day | 3
  Month 1: Frequency of symptoms: All day | 1
  Month 1: Frequency of symptoms: 24 hours a day | 1
  Month 1: Frequency of symptoms: Response missing | 7
  Month 1: Impact of symptoms on activities: Not applicable | 19
  Month 1: Impact of symptoms on activities: prohibits certain activities | 3
  Month 1: Impact of symptoms on activities: temporary stop of activities | 2
  Month 1: Impact of symptoms on activities: continue activities | 1
  Month 1: Impact of symptoms on activities: response missing | 7
  Month 1: pre- and post-operative pain: Not applicable | 21
  Month 1: pre- and post-operative pain: post-operative discomfort < Hernia discomfort | 3
  Month 1: pre- and post-operative pain: Post-operative discomfort > Hernia discomfort | 1
  Month 1: pre- and post-operative pain: response missing | 7
  Month 12: Location of symptoms: Not applicable: number analyzed (Participants) | 16
  Month 12: Location of symptoms: Not applicable | 15
  Month 12: Location of symptoms: Elsewhere: number analyzed (Participants) | 16
  Month 12: Location of symptoms: Elsewhere | 1
  Month 12: Timing of symptoms: Not applicable: number analyzed (Participants) | 16
  Month 12: Timing of symptoms: Not applicable | 15
  Month 12: Timing of symptoms: After exertion or end of day: number analyzed (Participants) | 16
  Month 12: Timing of symptoms: After exertion or end of day | 1
  Month 12: Frequency of symptoms: Not applicable: number analyzed (Participants) | 16
  Month 12: Frequency of symptoms: Not applicable | 15
  Month 12: Frequency of symptoms: Often during day: number analyzed (Participants) | 16
  Month 12: Frequency of symptoms: Often during day | 1
  Month 12: Impact of symptoms on activities: Not applicable: number analyzed (Participants) | 16
  Month 12: Impact of symptoms on activities: Not applicable | 15
  Month 12: Impact of symptoms on activities: Prohibits certain activities: number analyzed (Participants) | 16
  Month 12: Impact of symptoms on activities: Prohibits certain activities | 1
  Month 12: pre- and post-operative pain: Not applicable: number analyzed (Participants) | 16
  Month 12: pre- and post-operative pain: Not applicable | 14
  Month 12: pre- and post-operative pain: Post-operative discomfort > Hernia discomfort: number analyzed (Participants) | 16
  Month 12: pre- and post-operative pain: Post-operative discomfort > Hernia discomfort | 1
  Month 12: pre- and post-operative pain: Response missing: number analyzed (Participants) | 16
  Month 12: pre- and post-operative pain: Response missing | 1
  Month 24: Location of symptoms: Not applicable: number analyzed (Participants) | 4
  Month 24: Location of symptoms: Not applicable | 3
  Month 24: Location of symptoms: Bilateral: number analyzed (Participants) | 4
  Month 24: Location of symptoms: Bilateral | 1
  Month 24: Timing of symptoms: Not applicable: number analyzed (Participants) | 4
  Month 24: Timing of symptoms: Not applicable | 3
  Month 24: Timing of symptoms: Anytime: number analyzed (Participants) | 4
  Month 24: Timing of symptoms: Anytime | 1
  Month 24: Frequency of symptoms: Not applicable: number analyzed (Participants) | 4
  Month 24: Frequency of symptoms: Not applicable | 4
  Month 24: Impact of symptoms on activities: Not applicable: number analyzed (Participants) | 4
  Month 24: Impact of symptoms on activities: Not applicable | 3
  Month 24: Impact of symptoms on activities: Does not disrupt activities: number analyzed (Participants) | 4
  Month 24: Impact of symptoms on activities: Does not disrupt activities | 1
  Month 24: pre- and post-operative pain: Not applicable: number analyzed (Participants) | 4
  Month 24: pre- and post-operative pain: Not applicable | 3
  Month 24: pre- and post-operative pain: post-operative discomfort < Hernia discomfort: number analyzed (Participants) | 4
  Month 24: pre- and post-operative pain: post-operative discomfort < Hernia discomfort | 1
  Month 12: Perception of structure of abdominal wall: Solid: number analyzed (Participants) | 16
  Month 12: Perception of structure of abdominal wall: Solid | 16
  Month 12: Perception of lump in abdominal wall: No: number analyzed (Participants) | 16
  Month 12: Perception of lump in abdominal wall: No | 15
  Month 12: Perception of lump in abdominal wall: Elsewhere: number analyzed (Participants) | 16
  Month 12: Perception of lump in abdominal wall: Elsewhere | 1
  Month 24: Perception of structure of abdominal wall: Solid: number analyzed (Participants) | 4
  Month 24: Perception of structure of abdominal wall: Solid | 4
  Month 24: Perception of lump in abdominal wall: No: number analyzed (Participants) | 4
  Month 24: Perception of lump in abdominal wall: No | 4

6. Secondary Outcome: Surgeon Satisfaction
Description: Surgeon satisfaction on mesh ease of use and manipulability.
Time Frame: Day 0
Population: Surgeons who placed the ProGrip Self-Gripping Polyester Mesh during midline laparotomy procedures.
Measure: Number; unit: surgeons
Groups:
- Surgeons Placing ProGrip™ Self-Gripping Polyester Mesh: Survey administered to surgeons regarding ProGrip™ Self-Gripping Polyester Mesh
Arm/Group | Surgeons Placing ProGrip™ Self-Gripping Polyester Mesh
Number analyzed (Participants) | 26
surgeons
  Flexibility of the Mesh : Satisfactory | 25
  Flexibility of the Mesh : Not Stated | 1
  Cuttable : Satisfactory | 24
  Cuttable : Not Stated | 2
  Mesh shape memory : Satisfactory | 24
  Mesh shape memory : Unsatisfactory | 1
  Mesh shape memory : Not Stated | 1
  Mesh placement - adhesion to the wall: number analyzed (Participants) | 25
  Mesh placement - adhesion to the wall | 17
  Mesh placement - absence of laying direction: number analyzed (Participants) | 25
  Mesh placement - absence of laying direction | 8
  Mesh placement - shape memory: number analyzed (Participants) | 25
  Mesh placement - shape memory | 5
  Mesh placement - transparency: number analyzed (Participants) | 25
  Mesh placement - transparency | 8
  Mesh placement - easy to reposition: number analyzed (Participants) | 25
  Mesh placement - easy to reposition | 12

7. Secondary Outcome: Patient Satisfaction
Description: The Club Hernie Patient Satisfaction Survey is used to determine how satisfied a subject is with the mesh placement.
Time Frame: Month 12, Month 24
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Patients Treated With ProGrip Self-Gripping Polyester Mesh: Gripping Polyester Mesh: ProGrip™ Self-Gripping Polyester Mesh: All subjects enrolled receiving the ProGrip™ Self-Gripping Polyester Mesh
Arm/Group | Patients Treated With ProGrip Self-Gripping Polyester Mesh: Gripping Polyester Mesh
Number analyzed (Participants) | 16
participants
  Month 12: Repeat Procedure Performed = No | 14
  Month 12: Repeat Procedure Performed = Response Missing | 2
  Month 12: Strength of abdominal wall = Excellent | 5
  Month 12: Strength of abdominal wall = Good | 5
  Month 12: Strength of abdominal wall = Moderate | 1
  Month 12: Strength of abdominal wall = Poor | 1
  Month 12: Strength of abdominal wall = response missing | 4
  Month 24: Repeat Procedure Performed = No: number analyzed (Participants) | 4
  Month 24: Repeat Procedure Performed = No | 4
  Month 24: Strength of abdominal wall = Excellent: number analyzed (Participants) | 4
  Month 24: Strength of abdominal wall = Excellent | 1
  Month 24: Strength of abdominal wall = Good: number analyzed (Participants) | 4
  Month 24: Strength of abdominal wall = Good | 3
  Month 24: Strength of abdominal wall = Poor: number analyzed (Participants) | 4
  Month 24: Strength of abdominal wall = Poor | 0

8. Secondary Outcome: Surgeon Satisfaction
Description: Time to position the mesh
Time Frame: Day 0
Population: Surgeons who placed the ProGrip Self-Gripping Polyester Mesh during midline laparotomy procedures.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Surgeons Placing ProGrip™ Self-Gripping Polyester Mesh
Number analyzed (Participants) | 20
minutes | 8.0 (6.34)

ADVERSE EVENTS:
Time Frame: surgery to the 24-month visit
Groups:
- Patients Treated With ProGrip™ Self-Gripping Polyester Mesh: ProGrip™ Self-Gripping Polyester Mesh: All subjects enrolled will receive the ProGrip™ Self-Gripping Polyester Mesh
Arm/Group | Patients Treated With ProGrip™ Self-Gripping Polyester Mesh
All-Cause Mortality (participants affected / at risk) | 2/32
Serious Adverse Events (participants affected / at risk) | 10/32
Other Adverse Events (participants affected / at risk) | 17/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Treated With ProGrip™ Self-Gripping Polyester Mesh (N=32)
Arrhythmia (Cardiac disorders) | 1 (1)
Gastrointestinal fistula (Gastrointestinal disorders) | 1 (1)
Gastrointestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Swelling (General disorders) | 1 (1)
Escherichia infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 1 (1)
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 1 (1)
Wound evisceration (Injury, poisoning and procedural complications) | 2 (2)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Small intestinal resection (Surgical and medical procedures) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Shock (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Treated With ProGrip™ Self-Gripping Polyester Mesh (N=32)
Arrhythmia (Cardiac disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Fistula of small intestine (Gastrointestinal disorders) | 1 (1)
Gastrointestinal fistula (Gastrointestinal disorders) | 1 (1)
Gastrointestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Steatorrhoea (Gastrointestinal disorders) | 1 (1)
Inflammation (General disorders) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Swelling (General disorders) | 1 (1)
Escherichia infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Vascular device infection (Infections and infestations) | 1 (1)
Anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 2 (2)
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 1 (1)
Wound evisceration (Injury, poisoning and procedural complications) | 2 (2)
Investigation (Investigations) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Small intestinal resection (Surgical and medical procedures) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Shock (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to unsuccessful attempts to limit inclusion of complex patients with severe and multiple comorbidities at high risk of surgical complications that are not related to study device, and due to limited sample size, it was no longer feasible to clinically interpret the evidence from this study, leading to its early termination. Consequently, most planned analyses were not able to be performed. Limited data were collected, which affected the primary and secondary endpoint analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/62/NCT03912662/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/62/NCT03912662/SAP_001.pdf